CLINICAL TRIAL: NCT04069793
Title: Determining the Functional Importance of a Powered Multifunction Wrist
Brief Title: Functional Importance of a Powered Multifunction Wrist Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Levi Hargrove, Director of the Center for Bionic Medicine, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STU00206531; 5R01HD094861-02 (NIH)
Record Dates: First submitted 2019-08-09; First posted 2019-08-28 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Upper Limb Amputation at the Hand; Upper Limb Amputation at the Wrist; Amputation; Amputation; Traumatic, Limb
Keywords: Transradial Amputee

STUDY DESIGN:
Intervention Model Description: Study Design includes using the subjects to complete both aims in a balanced randomized cross-over study.
  Using blocked randomization, which will be achieve using a simple randomization script written in
  Matlab. The two study conditions that will be analyzed are:
  Condition A-a single DOF terminal device with a 1-DOF (rotation) wrist Condition B-a single DOF terminal device with a 2-DOF (rotation + flexion/extension) wrist
  Condition A is the control condition in this project as it represents the state-of-the-art in clinical care. Condition B is the experimental arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home Trial Condition A (Active Comparator): Subject will use a pattern recognition controlled prosthesis that includes a powered wrist rotation, passive wrist flexion/extension, and a single DOF powered hand.
  Interventions: Device: Commercially available device
- Home Trial Condition B (Experimental): Subject will use at pattern recognition controlled prosthesis that includes a powered wrist rotation, powered flexion/extension and a single DOF powered hand.
  Interventions: Device: Non FDA registered device

INTERVENTIONS:
Device: Commercially available device — A commercially available and registered with the FDA prosthesis equipped with a powered single-degree of freedom wrist and powered hand.
  Arms: Home Trial Condition A
Device: Non FDA registered device — An experimental, non FDA registered prosthesis equipped with a multi function wrist and a powered hand.
  Arms: Home Trial Condition B

SUMMARY:
The focus of this study is to conduct a clinical study in individuals with transradial amputations to compare function using a 1-DOF or 2-DOF wrist. All prostheses will be attached to a single DOF Otto Bock hand and controlled using a pattern recognition system equivalent to the Coapt system. This study will enable the investigator to quantify the relative functional value of powered wrist flexion during both in-laboratory testing and home use. In addition, the investigators will address the effectiveness of different hand-wrist combinations to enhance patient-centered clinical decision making.

DETAILED DESCRIPTION:
The primary objective of this project is to evaluate the functional importance of a multi function wrist compared to a single degree of freedom wrist. This will be accomplished through in laboratory testing and an 8-week home trial. The first aim will involve in-laboratory functional performance testing with a 1-DOF or a 2-DOF wrist and a one degree of freedom hand.

Changes in performance will be assessed with multiple outcome measures that include both quantitative and qualitative testing of prosthesis control and functional performance. The second aim will determine how a 2-DOF wrist impacts control and home use of a one degree of freedom hand. Subjects will compete an 8 week home based trial. Participants will be instructed to complete a written home log of activities and electronic logging usage data will also be collected for each experimental condition. The investigators hypothesize that adding a wrist flexion/extension module to a wrist rotation module and a single-DOF terminal device will provide significant improvements in function for transradial amputees.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-95
* A unilateral upper limb amputation or absence below the elbow
* English speaking

Exclusion Criteria:

* Significant new injury that would prevent use of a prosthesis: The ability to consistently wear a prosthesis and perform activities of daily living and specific performance tasks is necessary to evaluate the relative benefits of the interventions.
* Cognitive impairment sufficient to adversely affect understanding of or compliance with study requirements, ability to communicate experiences, or ability to give informed consent: The ability to understand and comply with requirements of the study is essential in order for the study to generate useable, reliable data. The ability to obtain relevant user feedback through questionnaires and informal discussion adds significant value to this study.
* Significant other comorbidity: Any other medical issues or injuries that would preclude completion of the study, use of the prostheses, or that would otherwise prevent acquisition of useable data by researchers

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Academy of Prosthetics and Orthotics ULPOM committee toolkit of outcome measures to record change of prosthetic performance | Baseline and 8 weeks for Condition A; Baseline and 8 weeks for Condition B
  Measuring the function of upper limb prostheses is challenging and requires multiple test formats. A toolkit of functional outcome tests recommend by the Academy of Prosthetics and Orthotics ULPOM committee will be used to measure functional effectiveness of prosthetic treatment will be used as the primary outcome measure. The outcome measures to evaluate prosthesis use includes both quantitative and qualitative testing of prosthesis control and functional performance.

SECONDARY OUTCOMES:
SHAP: Southampton Hand Assessment Procedure; a clinically validated hand function test to assess the effectiveness of upper limb prostheses. | Baseline and 8 weeks for Condition A; Baseline and 8 weeks for Condition B
  An objective test of unilateral hand function that can be used to evaluate functionality of passive, mechanical, or myoelectric hands without bias to type [31]. Movement of abstract objects (classified into six prehension patterns) and activities of daily living are timed by the subject. Scores are compared to a normalized, able-bodied control score of 100.
Modified Box and Blocks Test of Manual Dexterity | Baseline and 8 weeks for Condition A; Baseline and 8 weeks for Condition B
  A timed test that evaluates gross manual dexterity. Small (1-inch) blocks are moved one at a time from one side of a box to the other over a wooden partition. The final score is the number of blocks transferred in 1 minute, typically averaged over three trials. For this test, only opening and closing of the terminal device is required, although subjects with transradial amputations do typically use compensatory movements. It is possible that a 2-DOF wrist may move inadvertently and impair performance on this task. As a result, we would view either an improvement or no change in this score to be a positive finding.
Jebsen-Taylor Hand Function Test | Baseline and 8 weeks for Condition A; Baseline and 8 weeks for Condition B
  A standardized test of manual dexterity that evaluates hand function during performance of seven hand-related tasks using common items such as cards, cans, paper clips, and coins [32]. Subjects are evaluated by the time required to complete each task
Assessment of Capacity for Myoelectric Control (ACMC) | Baseline and 8 weeks for Condition A; Baseline and 8 weeks for Condition B
  An observational assessment tool that measures the subject's ability to control a myoelectric hand. The ability to control gripping, holding, releasing, and coordinating 30 items is scored on a 4-point capability scale. The prosthetic hand is used in an active assist or passive support role. Rasch analysis is used to convert capability ratings to a single measure of each subject's functional ability. Both Ms Turner and Dr. Miller are trained to complete this assessment.
Orthotics and Prosthetics User Survey - Upper Extremity Function Status | Baseline and 8 weeks for Condition A; Baseline and 8 weeks for Condition B
  A 19- item, self-reported measure of an individual's ability to perform self-care and upper limb-based daily living tasks (e.g. button shirt, tie shoelaces) using a 5-point scale [35]. Rasch analysis of the questionnaire ratings is used to calculate an overall measure of each subject's functional ability.
Patient Specific Functional Scale | Baseline and 8 weeks for Condition A; Baseline and 8 weeks for Condition B
  A questionnaire that asks patients to list up to five tasks they have difficulty with and rate the difficulty on an 11-point numerical scale [36]. Difficulty ratings can be averaged for each participant.
Clothespin Relocation Test | Baseline and 8 weeks for Condition A; Baseline and 8 weeks for Condition B
  A test of prosthetic function that requires the user to move three clothespins from a vertical bar to a horizontal bar (thereby requiring use of the elbow, terminal device, and wrist rotator). This test has been in use by CBM as a measure of prosthesis function for over a decade.
Virtual Testing: Target Achievement Control Test | 2 days
  For the TAC Test, participants must move the virtual hand into a target posture and hold it there for a preset period of time. The TAC Test can require movement of from one to all available degrees of freedom (e.g. hand grasp plus wrist motion). Results are measured in terms of classification accuracy, completion rate, completion time, and path efficiency. This test will be used to ensure that subjects have satisfactory PR control over all DOFs prior to starting their home trial.

CONTACTS AND LOCATIONS:
Overall Officials: Levi Hargrove, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No